CLINICAL TRIAL: NCT01132560
Title: A Correlative Science Study for ECOG E5194
Brief Title: Biomarkers in Tissue Samples From Patients With Ductal Breast Carcinoma in Situ
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000671157; ECOG-E5194T1
Record Dates: First submitted 2010-05-26; First posted 2010-05-28 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating | interventions — Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: RNA analysis
Genetic: gene expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is studying biomarkers in tissue samples from patients with ductal breast carcinoma in situ.

DETAILED DESCRIPTION:
OBJECTIVES:

* To validate the prognostic utility of a new ductal breast carcinoma in situ (DCIS) genomic score and the Oncotype DX Recurrence Score® assay in tissue samples from patients with DCIS enrolled on clinical trial ECOG-E5194.

OUTLINE: RNA extracted from archived tissue samples are analyzed for gene expression profile by Oncotype DX Recurrence Score® assay (a reverse transcriptase-PCR-based assay).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of ductal breast carcinoma in situ
* Enrolled on clinical trial ECOG-E5194

  * Local surgery without radiotherapy
  * Treated or not treated with tamoxifen
* Available tissue samples
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patient enrolled on E5194
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2010-03-05 (Actual); Primary Completion 2010-04-05 (Actual); Study Completion 2010-04-05 (Actual)

PRIMARY OUTCOMES:
Ipsilateral local failure (first event of invasive or DCIS recurrence) | 1 month

SECONDARY OUTCOMES:
Contralateral breast cancer (invasive or DCIS) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J. Solin, MD, FACR, Principal Investigator — Abramson Cancer Center at Penn Medicine